CLINICAL TRIAL: NCT03244930
Title: Low Dose Plerixafor Plus G-CSF Efficiency in Mobilizing Stem Cells From Lymphoma and Myeloma Patients for Autologous Peripheral Blood Transplantation
Brief Title: Low Dose Plerixafor Plus G-CSF in Mobilizing Stem Cells for Autologous Peripheral Blood Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Hematology division chief, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE17-00007
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Hodgkin; Myeloma; Stem Cell Transplant Complications
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Neoplasms, Plasma Cell | interventions — plerixafor

STUDY DESIGN:
Intervention Model Description: Prospective, open-labeled, single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Plerixafor 0.12 mg/kg SC will be administered in the evening, 11 hours prior to initiation of apheresis. G-CSF will be administered in the morning at 10 mcg/kg SC for 4 days prior to apheresis.
  Interventions: Drug: Plerixafor 0.12 mg/kg

INTERVENTIONS:
Drug: Plerixafor 0.12 mg/kg — Subcutaneously G-CSF 10 mg/kg for 4 days. At day four SC plerixafor 0.12 mg/kg as a single dose 11 hours prior to initiation of aphaeresis.
  Other Names: mozobil

SUMMARY:
Plerixafor, is added to mobilizing chemotherapy and G-CSF to overcome poor stem cell mobilization. We want to demonstrate that half of the commonly prescribed dose can be safely administered once as a single dose in first attempt leading to apheresis yields of >2 x 106 CD34+ cells/kg body weight.

DETAILED DESCRIPTION:
Plerixafor, is added to mobilizing chemotherapy and G-CSF to overcome poor stem cell mobilization. Consecutive patients in autologous transplant protocol will receive mobilization consisted of daily subcutaneously G-CSF 10 mg/kg for 4 days and plerixafor 0.12 mg/kg as a single dose 11 hours prior to initiation of apheresis. HSC collection was performed with a Cobe Spectra® or Spectra Optia® apheresis system. The planned target blood volume to be processed will be 4-fold total blood volume calculated according to patients' weight and size. Peripheral blood CD34+ counts will be analyzed using flow cytometry. For each ASCT, we aimed for target yields of at least 2 x 106 CD34+cells/kg. Toxicities and engraftment will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Candidates planned for an autologous haematopoietic stem cell transplantation without previous mobilization attempts with chemotherapy.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
3. WBC count ≥2.5x109/L.
4. Absolute neutrophil count ≥1.5x109/L.
5. Platelet count ≥100x109/L

Exclusion Criteria:

1. Prior allogeneic or autologous transplantation.
2. Pregnant women.
3. Acute infection (febrile, i.e. temperature > 38C) within 24 hours prior to dosing or antibiotic therapy within 7 days prior to the first dose of GCSF.
4. Positive serology for hepatitis B or C or HIV.
5. Left ventricular ejection fraction < 40%
6. AST ALT >2.5x or Creatinine >2 md/dL

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-05-10 (Estimated); Study Completion 2018-06-10 (Estimated)

PRIMARY OUTCOMES:
Harvest of of at least 2 x106 CD34+/kg | 5 days
  percentage of patients with a target yields of at least 2 x 106 CD34+ cells/kg in one single aphaeresis procedure.

SECONDARY OUTCOMES:
Time to engraftment | 100 days
  Engraftment defined as 3 consecutive days of neutrophil counts higher than 0.5 x 103/mcl
Rate of patients reaching a peripheral blood precount higher than 20 cells/μL | 5 days
  Rate of patients reaching a peripheral blood precount higher than 20 cells/μL

CONTACTS AND LOCATIONS:
Overall Officials: David Gomez Almaguer, md, Study Director — Servicio de Hematología Hospital Universitario "Dr. José Eleuterio Gonzalez"
Locations (1):
- Servicio de Hematología Hospital Universitario "Dr. José Eleuterio Gonzalez", Universidad Autónoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Result] DiPersio JF, Micallef IN, Stiff PJ, Bolwell BJ, Maziarz RT, Jacobsen E, Nademanee A, McCarty J, Bridger G, Calandra G; 3101 Investigators. Phase III prospective randomized double-blind placebo-controlled trial of plerixafor plus granulocyte colony-stimulating factor compared with placebo plus granulocyte colony-stimulating factor for autologous stem-cell mobilization and transplantation for patients with non-Hodgkin's lymphoma. J Clin Oncol. 2009 Oct 1;27(28):4767-73. doi: 10.1200/JCO.2008.20.7209. Epub 2009 Aug 31. PMID 19720922
- [Result] Flomenberg N, Comenzo RL, Badel K, Calandra G. Plerixafor (Mozobil) alone to mobilize hematopoietic stem cells from multiple myeloma patients for autologous transplantation. Biol Blood Marrow Transplant. 2010 May;16(5):695-700. doi: 10.1016/j.bbmt.2009.12.538. Epub 2010 Jan 11. PMID 20067838
- [Result] Brave M, Farrell A, Ching Lin S, Ocheltree T, Pope Miksinski S, Lee SL, Saber H, Fourie J, Tornoe C, Booth B, Yuan W, He K, Justice R, Pazdur R. FDA review summary: Mozobil in combination with granulocyte colony-stimulating factor to mobilize hematopoietic stem cells to the peripheral blood for collection and subsequent autologous transplantation. Oncology. 2010;78(3-4):282-8. doi: 10.1159/000315736. Epub 2010 Jun 8. PMID 20530974
- [Result] Haverkos BM, Huang Y, Elder P, O'Donnell L, Scholl D, Whittaker B, Vasu S, Penza S, Andritsos LA, Devine SM, Jaglowski SM. A single center's experience using four different front line mobilization strategies in lymphoma patients planned to undergo autologous hematopoietic cell transplantation. Bone Marrow Transplant. 2017 Apr;52(4):561-566. doi: 10.1038/bmt.2016.304. Epub 2017 Jan 9. PMID 28067870
- [Derived] Gutierrez-Aguirre CH, Alvarado-Navarro DM, Palomares-Leal A, Mejia-Jaramillo G, Salazar-Riojas R, Leon AG, Colunga-Pedraza PR, Sotomayor-Duque G, Jaime-Perez JC, Cantu-Rodriguez OG, Del Carmen Tarin-Arzaga L, Flores-Jimenez JA, Gomez-Almaguer D. Reduced-dose plerixafor as a mobilization strategy in autologous hematopoietic cell transplantation: a proof of concept study. Transfusion. 2019 Dec;59(12):3721-3726. doi: 10.1111/trf.15547. Epub 2019 Oct 16. PMID 31618456